CLINICAL TRIAL: NCT01219166
Title: Is Routine Cholecystectomy Reasonable in All Patients Receiving a Bypass Procedure: a Comparative Cohort Study
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Andreas Zerz, MD, Kantonal Hospital St. Gallen, Department of Visceral Surgery
Other Study IDs: EKSG10/140/U
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-10

CONDITIONS: Given Indication for Gastric Bypass Procedure
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- laparoscopic Roux-en-Y-gastric-bypass without cholecystectomy
- laparoscopic Roux-en-Y-gastric baypass with cholecystectomy
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Laparoscopic Cholecystectomy
  Groups: laparoscopic Roux-en-Y-gastric baypass with cholecystectomy

SUMMARY:
Gallbladder management in bariatric surgery is controversially discussed. While some surgeons advocate routine prophylactic cholecystectomy (CCE) during Roux-en-Y gastric bypass (RYGB) others advocate CCE only in patients with pathological gallbladder findings. The aim of this study was to evaluate the necessity of prophylactic CCE in patients receiving a laparoscopic RYGB.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received a laparoscopic Roux-en-Y-gastric bypass

Exclusion Criteria:

* previous CCE
* open gastric bypass procedure
* previous bariatric procedure other than gastric banding
* patients lost to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Given indication for laparoscopic Roux-en-Y-gastric bypass
Sampling Method: Non-Probability Sample
Enrollment: 437 (Estimated)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
biliary complications resulting from omitted prophylactic cholecystectomy | 5 years

SECONDARY OUTCOMES:
safety of concurrent cholecystectomy | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin Thurnheer, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Department of surgery, Sankt Gallen, Switzerland